CLINICAL TRIAL: NCT06067503
Title: Integrating Minimally Invasive Biomarkers of Estrogen Signaling to Detect Endocrine Therapy Resistance in Metastatic Invasive Lobular Breast Cancer
Brief Title: Biomarkers to Detect Endocrine Therapy Resistance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-1103; Protocol Version 10/2/2023 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); UW23076 (Other: OnCore ID)
Record Dates: First submitted 2023-09-19; First posted 2023-10-05 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Cancer; Breast Cancer; Lobular Breast Carcinoma
Keywords: Endocrine Therapy Resistance; circulating tumor cell; liquid biopsy
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Carcinoma, Lobular; Neoplastic Cells, Circulating | interventions — Liquid Biopsy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with ER/PR+ metastatic lobular breast cancer (LBC) (Experimental)
  Interventions: Drug: 18F-fluorofuranylnorprogesterone; Device: Liquid Biopsy; Device: Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Drug: 18F-fluorofuranylnorprogesterone — The dose of the investigational imaging agent, FFNP, is approximately 7 millicurie (mCi) (259 megabecquerels (MBq)), IV slow infusion over approximately two minutes followed by saline flush.
  Other Names: FFNP
Device: Liquid Biopsy — 20ml of whole blood will be collected into two Ethylenediaminetetraacetic acid (EDTA) tubes at each timepoint, CTCs are isolated using the microfluidic Versatile Exclusion-based Rare Sample Analysis (VERSA) platform that integrates CTC capture with RNA extraction on a single chip using Exclusion-Based Sample Preparation (ESP) technology
  Other Names: Circulating Tumor Cells (CTC)
Device: Positron Emission Tomography/Computed Tomography — FFNP drug in combination with PET/CT scans to image participant
  Other Names: PET/CT

SUMMARY:
This pilot observational study is being done to identify possible biomarkers of response to endocrine therapy in patients with ER/PR+ metastatic lobular breast cancer (LBC) starting new endocrine therapy. 18F-fluorofuranylnorprogesterone Positron Emission Tomography/Computed Tomography (FFNP-PET/CT) and liquid biopsies will be performed at baseline and after 4 weeks of treatment. Baseline levels and dynamic on-treatment changes in estrogen signaling as measured by FFNP-PET/CT and circulating tumor cell (CTC) liquid biopsy will be correlated with clinical response to endocrine therapy and progression-free survival in the above cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent
2. Individuals at least 18 years of age
3. Have biopsy-proven ER/PR-positive (defined as ER ≥1 percent and PR ≥1 percent by IHC) and HER2-negative advanced or metastatic LBC starting new standard of care endocrine therapy
4. Adequate organ function as indicated by standard laboratory tests (CBC, liver function tests or CMP) allowing for systemic breast cancer treatment per treating oncologist
5. Patients with evaluable bone-only disease that is lytic or mixed lytic-sclerotic are eligible
6. Willing to comply with all study procedures and be available for the duration of the study
7. Disease may be measurable by RECIST 1.1 criteria or non-measurable. Lesion size must be at least 1cm. If only bone lesions present, they should be lytic or mixed lytic-sclerotic. If only liver lesions present, patient is not eligible.

Exclusion Criteria:

1. Patients with active brain metastases
2. Patients with liver-only disease are not eligible due to high background liver activity related to the radiopharmaceutical's hepatobiliary route of elimination
3. Unable to lie flat during or tolerate PET/CT
4. Patients with a history of allergic reaction attributable to compounds of similar chemical or biologic composition to FFNP
5. Presence of liver failure as judged by patient's treating physician
6. Individuals who are pregnant, lactating, or planning on becoming pregnant during the study
7. Not suitable for study participation due to other reasons at the discretion of the investigators
8. Patients with progesterone-receptor negative disease defined as PR <1 percent by IHC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who have decreased FFNP uptake on PET/CT in response to endocrine therapy | baseline, 4 weeks
Number of Participants who have decrease in circulating tumor cell estrogen signaling in response to endocrine therapy | baseline, 4 weeks
  Baseline level and on-treatment CTC ESR1 and estrogen regulated gene expression will be evaluated as well as endocrine-resistance associated mutations including ESR1 (though rare in this patient population) and PGR.
Number of Participants who have a decrease in concentration of Circulating Tumor DNA in response to endocrine therapy | baseline, 4 weeks

SECONDARY OUTCOMES:
Progression Free Survival (PFS) for 6 months | up to 6 months
Correlation coefficients | up to 6 months
  Correlate baseline levels and dynamic on treatment changes in estrogen signaling as measured by FFNP-PET/CT and CTC liquid biopsy with clinical response to endocrine therapy and progression-free survival in patients with ER/PR+ metastatic LBC.
Adverse Events within 24 hours of FFNP infusion | a 24 hour period up to 7 days pre-treatment, a 24 hour period 4 weeks after the first infusion

CONTACTS AND LOCATIONS:
Overall Officials: Marina Sharifi, MD, PHD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers up to 7 years after the completion of the primary endpoint by contacting the University of Wisconsin Carbone Cancer Center (UWCCC)
Time Frame: up to 7 years after the completion of the primary endpoint
Access Criteria: UWCCC Cancer Connect: clinicaltrials@cancer.wisc.edu